CLINICAL TRIAL: NCT04749953
Title: Maxillary Sinus Floor Augmentation With Autogenous Bone Graft Alone or in Combination With Symbios Biphasic Bone Graft Material or Symbios Xenograft Granules. A Randomized Controlled Trial
Brief Title: Maxillary Sinus Floor Augmentation With Different Grafting Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Starch-Jensen, Clinical Professor, chief surgeon, DDS, PhD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Thomas Starch-Jensen1
Record Dates: First submitted 2021-01-21; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Survival, Prosthesis; Peri-Implantitis; Patient Satisfaction
Keywords: Alveolar ridge augmentation; Maxillary sinus floor elevation; Patient-reported outcome measures; Dental implants; Biomaterials
MeSH Terms: conditions — Prosthesis Failure; Peri-Implantitis; Patient Satisfaction | interventions — Sinus Floor Augmentation

STUDY DESIGN:
Intervention Model Description: A single-blinded randomized controlled study. No drug or device is tested. Different grafting materials for bone augmentation is compared. Autogenous bone graft is golden standard, which is compared with two different mixtures of alternative grafting materials.
Who Masked: Participant
Masking Description: Patients are blinded to the used grafting material.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autogenous bone graft alone (Active Comparator): Maxillary sinus floor augmentation with particulated autogenous bone graft alone from the zygomatic buttress area and simultaneously implant placement
  Interventions: Procedure: Maxillary sinus floor augmentation
- Mixture of 50% autogenous bone graft and 50% Symbios biphasic biomaterial (Experimental): Maxillary sinus floor augmentation with a mixture of 50% particulated autogenous bone graft from the zygomatic buttress area and 50% Symbios biphasic bone graft material (Biomaterial, 1.0 mm to 2.0 mm) with simultaneously implant placementand
  Interventions: Procedure: Maxillary sinus floor augmentation
- Mixture of 50% autogenous bone graft and 50% Symbios xenograft granules (Experimental): Maxillary sinus floor augmentation with a mixture of 50% particulated autogenous bone graft from the zygomatic buttress area and 50% Symbios xenograft granules (Biomaterial, 1.0 mm to 2.0 mm) with simultaneously implant placement
  Interventions: Procedure: Maxillary sinus floor augmentation

INTERVENTIONS:
Procedure: Maxillary sinus floor augmentation — The sinus membrane of the maxillary sinus is elevated to create a space for the grafting material and placement of dental implants in the posterior maxilla

SUMMARY:
Implant placement in the posterior maxilla is compromised due to atrophy of the alveolar process and maxillary sinus pneumatisation. Bone augmentation is frequently necessary before or in conjunction with implant placement. The most commonly used method to augment the posterior maxillary involves maxillary sinus floor augmentation (MSFA) with autogenous bone graft or bone substitute. Autogenous bone graft harvesting is associated with risk of donor site morbidity and unpredictable resorption of graft. Thus, bone substitutes alone or in combination with autogenous bone are used increasingly to simplify the surgical procedure.

Symbios biphasic biomaterial is a resorbable inorganic bone forming material derived from red algae consisting of 20% hydroxylapatite and 80% β-tricalciumphosphate with osteoconductive properties. Histologic and radiographic examinations indicate that β-tricalciumphosphate is slowly resorbed and replaced with bone. MSFA with β-tricalciumphosphate alone or in combination with autogenous bone or other bone substitutes have demonstrated high implant survival and new bone.

Symbios xenograft granules is a porcine bone mineral with osteoconductive properties. Histologic and radiographic examinations indicate that xenograft is a non-resorbable graft material. MSFA with xenograft alone or in combination with autogenous bone have shown high implant survival and new bone.

The objective is to test the H0-hypothesis of no difference in implant outcome after MSFA with autogenous bone graft or in combination with Symbios biphasic biomaterial or Symbios xenograft. 60 consecutively healthy patients with a missing posterior maxillary tooth/teeth will be randomly allocated to: 1) MSFA with autogenous bone graft, 2) MSFA with mixture of 50% autogenous bone graft and 50% Symbios biphasic biomaterial 3) MSFA with mixture of 50% autogenous bone graft and 50% Symbios xenograft. Implants will be inserted simultaneously with MSFA. Clinical and/or radiographical evaluation using periapical radiographs and Cone Beam Computer Tomography will be performed preoperatively, immediate postoperatively, before abutment connection, after prosthetic rehabilitation, and after one year to assess the treatment outcome and volumetric changes of the augmented area. Outcome include survival of suprastructures and implants, volumetric stability of graft, peri-implant marginal bone level, oral health related quality of life, and complications.

DETAILED DESCRIPTION:
Maxillary sinus floor augmentation (MSFA) is the most frequently used method to enhance the alveolar bone of the posterior maxilla before or in conjunction with implant placement. Autogenous bone is considered as the preferred graft material due to its osteoinductive, osteogenic and osteoconductive characteristics. However, autogenous bone grafts is associated with risk of donor site morbidity and unpredictable graft resorption. Hence, various bone substitutes are used increasingly to simplify the surgical procedure by diminishing the need for bone harvesting. From a clinical and patient perspective, it would be an advantage, if autogenous bone grafts could partially or totally be replaced with bone substitutes.

Symbios xenograft is a new porcine bone mineral characterized as an anorganic bone matrix with an interconnecting macro- and microscopic pore structure that supports formation and in-growth of new bone. Porcine xenograft have previously been used for various augmentation procedures disclosing new bone formation. Studies comparing autogenous bone graft with porcine bone alone or a mixture of autogenous bone and porcine bone have demonstrated high implant survival and new bone.

Synthetic biomaterials including calcium phosphate, calcium sulphate, polymers and bioactive glass represent a large group of inorganic diverse biomaterials with variating structures, chemical composition and physical properties. Symbios biphasic biomaterials is a resorbable inorganic bone forming material derived from red algae consisting of 20% hydroxylapatite and 80% β-tricalciumphosphate. Studies assessing MSFA with β-tricalciumphosphate have demonstrated that it is a safe grafting material with osteoconductive properties. Histologic and radiographic examinations indicate that β-tricalciumphosphate is slowly resorbed and replaced with bone. MSFA with β-tricalciumphosphate alone or in combination with autogenous bone or other bone substitutes have demonstrated high implant survival and new bone.

The study purpose is to increase our knowledge about MSFA with autogenous bone alone or in combination with Symbios biphasic biomaterials or Symbios xenograft granules and to simplified the procedure. Evaluation will include survival of suprastructures and implants, peri-implant marginal bone level, volumetrical stability of the graft and complications after an observation period of one year. Furthermore, oral health related quality of life, using OHIP-14 self-administrated and patient satisfaction using visual analogue scales (VAS), will be evaluated.

The objective is to test the H0 hypothesis of no differences in 1) Survival of suprastructures and implants, 2) Volumetrical stability of the graft, 3)Peri-implant marginal bone level, 4) Implantat stability quotient, 5) Patient-reported outcome measures, and 6) Biologic and technical complications.

Materials and methods Study population 60 consecutively healthy patients with a missing posterior maxillary tooth will be included and randomly allocated to: 1) MSFA with autogenous bone graft alone (control group), 2) mixture of 50% autogenous bone graft and 50% Symbios biphasic biomaterial (test group I), and 3) mixture of 50% autogenous bone and 50% Symbios xenograft (test group II). The study will be conducted at the Departments of Oral and Maxillofacial Surgery, Aalborg University Hospital, Denmark and Oral and Maxillofacial Surgery and Oral Medicine, Malmö University, Malmö, Sweden.

Patients will be included to the study by using a Facebook posting through the University's Facebook page, the local dental association website or patients that are referred to the Departments for treatment of one or more missing teeth in the posterior maxilla. All patients will be offered participation in the study, if they meet the inclusion criteria. Prior to patients' first visit, they will receive a notice informing about their rights and informed consent form will be signed.

Inclusion criteria involves 1) >20 years, 2) Missing one or more posterior maxillary teeth, 3) Residual bone height of the maxillary alveolar process between 3 to 7 mm, 4) Width of the alveolar process ≥6.5 mm and, 5) Mandibular occluding teeth. Exclusion criteria involves 1) Contraindications to implant therapy, 2) Full mouth plaque score >25%, 3) Progressive marginal periodontitis, 4) Acute infection in the area intended for implant placement, 5)Parafunction, bruxism, or clenching, 6) Psychiatric problems or unrealistic expectations, 7) Heavy tobacco use, define as >10 cigarettes per day, and 8)Pregnancy.

The study is approved by the local ethical Committee on Health Research and the Danish Data Protection Agency and The Ethical Review Board in Lund, Sweden' and will be performed according to the Declaration of Helsinki on clinical research. All patients will be given verbal and written information about the study at a clinical visit prior to surgery. Written informed consent is mandatory for inclusion in the study and will be obtained by the investigators.

The initial examination of the patient will include 1) Clinical examination and screening of the parodontal health, 2) Radiographical examination of the residual alveolar bone height based on CBCT and Orthopantomography, and 3) Patient will fill out the OHIP-14 questionnaire.

The surgical procedure will be performed in local anesthesia. Implant installation and fabrication of the subsequently prosthetic solution will be performed according to manufacturer's recommendations. The maxillary sinus wall is exposed by an intraoral marginal incision from tuber maxillae to the first premolar with a vertical releasing incision. A 1 x 1 cm window to the maxillary sinus is created with metal and diamond burrs maintaining an intact Schneiderian membrane. The Schneiderian membrane is elevated from the sinus floor as well as the lateral sinus wall and displaced dorsocranially with blunt dissector. An implant bed is successively prepared on the top of the alveolar crest following manufactory's recommendations at 1500 rpm. A straight implant (ASTRA TECH Implant System EV 3.6, 4.2 or 4.8, 13 mm) is inserted with a cover screw. The implant stability quotient is measured for all inserted implants. A sealed randomization envelope is opened in order to allocate the patient to: 1) MSFA with particulated autogenous bone graft alone (control group), 2) a mixture of 50% particulated autogenous bone graft and 50% Symbios biphasic bone graft material (1.0 mm to 2.0 mm) (test group I), 3) a mixture of 50% particulated autogenous bone graft and 50% Symbios xenograft granules (1.0 mm to 2.0 mm) (test group II). The autogenous bone graft is harvested with a curved SafeScraper from the zygomatic buttress area. Specially prepared stainless steel cups (0.5 cm3 and 1 cm3) are used to estimate 1 cm3 of graft material for each inserted implant. The graft material will be soaked in autogenous blood from the surgical site until use. The sinus around the implant is packed with 1 cm3 graft material. The created window to the maxillary sinus is covered by a Symbios Collagen Membrane 15 x 20 mm. Periosteum and mucosa are sutured with Vicryl 4-0. Minor perforations of sinus membrane will be covered with a Symbios Collagen Membrane. If the sinus membrane is largely perforated the procedure will be cancelled, and the patient will be withdrawn from the study. No provisional restoration is inserted during the healing period. After six months of healing, the inserted implants in the three treatment groups are exposed via a crestal incision. Mucosa and periosteum are elevated and the cover screw is removed. The implant stability quotient is measured for all inserted implants. The implant is rinsed with saline and a prefabricated healing abutment is placed. The implants are manually tested for mobility and osseointegration by percussion. Mucosa is adapted and sutured with Vicryl 4-0. The prosthetic restoration will be initiated three weeks after the healing abutment has been placed.

Prosthetic restoration will include an individualized abutment and a fixed restoration performed by experienced prosthodontists with extensive clinical experience with implant-based prosthetics.

Patients will be scheduled for a postoperative clinical examination at baseline, and one year after loading. The following parameters will be recorded at each visit 1) Plaque and gingival index, probing pocket depth, and probing attachment level, 2) Oral health related quality of life - OHIP-14 and 3) Patient satisfaction (VAS).

Radiographical evaluation will include seven sets of periapical radiographs and CBCT obtained preoperatively, immediately postoperatively, after abutment connection, at baseline and one year after loading. To provide blinding of the radiographical evaluation, the CBCT-scans are coded. Volumetrical changes of the grafts are estimated by point counting and the method described originally by Cavalieri. To obtain an equivalent starting point for the systematic uniform random sampling of the CBCT-scans images involving the maxillary sinus, all images from the neighboring teeth to the implant bed are selected. The first CBCT images after the distal surface of the anterior neighboring tooth is sampled randomly using a random number table for each maxillary sinus. Every second CBCT image is selected to ensure an equal mutual distance between the selected 5-10 images. The original outline of the maxillary sinus before implant installation is recorded and superimposed on the corresponding images. A point grid test system is superimposed at random on all images, allowing 100-200 points to hit the graft of each maxillary sinus. The numbers of intersections over the graft are counted on each selected image. Cavalieri volume estimation principle is used to estimate the total volume of the graft.

V = t x a(p) x ΣP

Where V is volume, t is the distance between the sampled images, a(p) is the area associated with each test point corrected for magnification and ΣP is the total number of points hitting the graft.

Peri-implant marginal bone changes are evaluated by linear measurements on digital periapical radiographs and will be done on radiographs obtained at implant placement, baseline, and one year after loading. The distance from the implant-abutment connection to the marginal bone level will be measured mesially and distally parallel with the long-axis of the implant.

Data management and analysis including calculation of descriptive statistics are done using STATA. A power calculation are based on differences in marginal bone level changes preformed in a previous study involving replacement of a single tooth with 2 different protocols of implant treatment. The calculation is based on the observed changes in marginal bone level from insertion of the implant to abutment connection (a change of 0.65 mm and a standard deviation of 0.65), 17 patients in each group reaches a power of 97% at the 5%-level. With 15% to cover drop-outs, each treatment group should include 20 patients. The statistical evaluation is performed by analysis of variance. Scheffe´s multiple comparison test is used post hoc to determine the relative effect of the various graft types. Level of significance is 0.05.

ELIGIBILITY:
Inclusion Criteria:

* >20 years
* Missing one or more posterior maxillary teeth
* Residual bone height of the maxillary alveolar process between 3 to 7 mm
* Width of the alveolar process ≥6.5 mm.
* Mandibular occluding teeth

Exclusion Criteria:

* Contraindications to implant therapy
* Full mouth plaque score >25%
* Progressive marginal periodontitis
* Acute infection in the area intended for implant placement
* Parafunction, bruxism, or clenching
* Psychiatric problems or unrealistic expectations
* Heavy tobacco use, define as >10 cigarettes per day
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Survival of suprastructures | One year of implant loading
  Loss of suprastructures is defined as a total loss because of a non-treatable mechanical/or biological complication
Survival of implants | One year of implant loading
  Loss of implants is defined as removal of a non-integrated implant, mobility of previously clinical osseointegrated implant, and removal of non-mobile implants due to progressive peri-implant marginal bone loss and infection

SECONDARY OUTCOMES:
Volumetric changes of the graft material | One year of implant loading
  Radiographic measurement of the augmented area
Peri-implant marginal bone level | One year of functional loading
  Radiographic assessment of the marginal bone loss around the implants
Patient-reported outcome measures | One year of functional implant loading
  Oral Health Impact Profile-14 (OHIP-14) questionnaire is used to assess oral health-related quality of life (OHRQoL). OHIP-14 is organized into seven dimensions including functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability and handicap. Two items are used to measure each dimension and consequently the questionnaire consists of 14 items. Response format is as follows: Very often = 4; Fairly often or many times = 3; Occasionally = 2; Hardly ever or nearly never = 1; Never/I don´t know = 0. OHIP-14 scale ranged from 0 to 56 and dimension score ranged from 0 to 8. Values of the 14 items and each dimension were summed to calculate the OHIP-14 severity score. Higher scores indicating poorer OHRQoL. Recovery is examined by a 100mm (0 = minimal to 100 = maximum) visual analogue scale assessing pain, social isolation, working isolation, eating ability, speaking ability and sleep impairment.
Complications | One year of functional implant loading
  Loss of implants or grafting material due to infection

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Data will be crypted and only referable for the primary investigator